CLINICAL TRIAL: NCT02741167
Title: Pathophysiology of Inflammation After Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: HIPEC 2015-0529
Record Dates: First submitted 2016-03-30; First posted 2016-04-18 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Peritoneal Cancer
Keywords: peritoneal surface malignancies; cytoreductive surgery; hyperthermic intraperitoneal chemotherapy
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRS and HIPEC: Patients subjected to cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) due to primary or secondary peritoneal malignancy
  Interventions: Procedure: CRS and HIPEC

INTERVENTIONS:
Procedure: CRS and HIPEC — During CRS, all visible peritoneal tumors are removed. Consequently micrometastasis are removed with hyperthermic intraperitoneal chemotherapy

SUMMARY:
The purpose of this study is to assess the dynamics of inflammatory parameters in presence or absence of infectious complications after cytoreductive surgery with hyperthermic intraperitoneal chemotherapy.

DETAILED DESCRIPTION:
Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy is the treatment of choice in patients with primary or secondary peritoneal surface malignancies. However the survival benefit is achieved at the cost of increased morbidity and mortality due to an extensive surgery and intraoperative chemo-therapy. Among complications infectious complications are the most common. The early diagnosis of a potential fatal infection is therefore crucial to ensure a good outcome in patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (more than 18 years) subjected to CRS and HIPEC due to peritoneal malignancy.
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* No primary or secondary peritoneal surface malignancy
* No CRS and HIPEC
* Pregnancy
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (more than 18 years) subjected to cytoreductive surgery (CRS) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) due to peritoneal malignancy at our institution.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
C reactive protein (CRP) mg/l, receiver operating characteristic (ROC) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kuno Lehmann, Md. PhD, Principal Investigator — Dr. Kuno Lehmann, Division of Visceral Surgery and Transplantation, University Hospital Zurich, Ramistrasse 100, 8091 Zurich, Switzerland
Locations (1):
- Division of Visceral Surgery and Transplantation , University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chua TC, Yan TD, Saxena A, Morris DL. Should the treatment of peritoneal carcinomatosis by cytoreductive surgery and hyperthermic intraperitoneal chemotherapy still be regarded as a highly morbid procedure?: a systematic review of morbidity and mortality. Ann Surg. 2009 Jun;249(6):900-7. doi: 10.1097/SLA.0b013e3181a45d86. PMID 19474692
- [Background] Roviello F, Caruso S, Marrelli D, Pedrazzani C, Neri A, De Stefano A, Pinto E. Treatment of peritoneal carcinomatosis with cytoreductive surgery and hyperthermic intraperitoneal chemotherapy: state of the art and future developments. Surg Oncol. 2011 Mar;20(1):e38-54. doi: 10.1016/j.suronc.2010.09.002. Epub 2010 Dec 15. PMID 20888755
- [Background] Klein HJ, Csordas A, Falk V, Slankamenac K, Rudiger A, Schonrath F, Rodriguez Cetina Biefer H, Starck CT, Graf R. Pancreatic stone protein predicts postoperative infection in cardiac surgery patients irrespective of cardiopulmonary bypass or surgical technique. PLoS One. 2015 Mar 20;10(3):e0120276. doi: 10.1371/journal.pone.0120276. eCollection 2015. PMID 25793700
- [Background] Younan R, Kusamura S, Baratti D, Cloutier AS, Deraco M. Morbidity, toxicity, and mortality classification systems in the local regional treatment of peritoneal surface malignancy. J Surg Oncol. 2008 Sep 15;98(4):253-7. doi: 10.1002/jso.21057. PMID 18726887
- [Background] Votanopoulos K, Ihemelandu C, Shen P, Stewart J, Russell G, Levine EA. A comparison of hematologic toxicity profiles after heated intraperitoneal chemotherapy with oxaliplatin and mitomycin C. J Surg Res. 2013 Jan;179(1):e133-9. doi: 10.1016/j.jss.2012.01.015. Epub 2012 Mar 10. PMID 22480844
- [Background] Sonnenberg EM, Reinke CE, Bartlett EK, Collier KT, Karakousis GC, Holena DN, Kelz RR. Wind, water, wound, walk--do the data deliver the dictum? J Surg Educ. 2015 Jan-Feb;72(1):164-9. doi: 10.1016/j.jsurg.2014.05.019. Epub 2014 Aug 12. PMID 25131719
- [Result] Lehmann K, Eshmuminov D, Slankamenac K, Kranzbuhler B, Clavien PA, Vonlanthen R, Gertsch P. Where Oncologic and Surgical Complication Scoring Systems Collide: Time for a New Consensus for CRS/HIPEC. World J Surg. 2016 May;40(5):1075-81. doi: 10.1007/s00268-015-3366-0. PMID 26669784
- [Result] Capone A, Valle M, Proietti F, Federici O, Garofalo A, Petrosillo N. Postoperative infections in cytoreductive surgery with hyperthermic intraperitoneal intraoperative chemotherapy for peritoneal carcinomatosis. J Surg Oncol. 2007 Nov 1;96(6):507-13. doi: 10.1002/jso.20837. PMID 17708508
- [Derived] Roth L, Eshmuminov D, Laminger F, Koppitsch C, Schneider M, Graf TR, Gupta A, Kober F, Roka S, Gertsch P, Lehmann K. Systemic inflammatory response after hyperthermic intraperitoneal chemotherapy (HIPEC): The perfusion protocol matters! Eur J Surg Oncol. 2019 Sep;45(9):1734-1739. doi: 10.1016/j.ejso.2019.03.036. Epub 2019 Mar 29. PMID 30954352